CLINICAL TRIAL: NCT02160431
Title: Investigating the Neuropsychological Profile of Youth With Obsessive Compulsive Disorder (OCD)
Brief Title: Neuropsychological Profiles of Pediatric Obsessive Compulsive Disorder (OCD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate funding
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Kevin D. Stark, Professor, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-004-0024
Record Dates: First submitted 2013-07-15; First posted 2014-06-10 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Obsessive Compulsive Disorder (OCD)
Keywords: Children; OCD; CBT; Neuropsychological profiles
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CBT for pediatric OCD (Experimental): Participants complete standard CBT for OCD
  Interventions: Behavioral: CBT for pediatric OCD

INTERVENTIONS:
Behavioral: CBT for pediatric OCD — Participants complete standard CBT for OCD as delivered in the POTS study .

SUMMARY:
The neuropsychological profiles of children treated with standard CBT for OCD are evaluated.

DETAILED DESCRIPTION:
The neuropsychological profiles of children treated with standard CBT for the treatment of OCD will be compared at pre-treatment and post-treatment. Children between the ages of 8 and 16 years who have a primary diagnosis of OCD will be participants. Treatment will last 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Children 8-16 years old who have a primary diagnosis of Obsessive Compulsive Disorder

Exclusion Criteria:

* Risk of suicidal or homicidal behavior
* Presence of another psychological disorder as the primary disorder
* Psychotic disorder, bipolar disorder, Pervasive Developmental Disorder, Thought Disorder, Uncontrolled ADHD, Eating Disorder, Substance Use Disorders, School refusal behavior characterized by missing more than 25% of days in most recent term, does not speak English, youth does not have at least one parent who speaks English

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2014-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Children's Yale Brown Obsessive Compulsive Scale measures change in severity of OCD symptoms from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Measures presence and severity of obsessions and compulsions.

SECONDARY OUTCOMES:
Anxiety Disorders Interview Schedule-Diagnostic and Statistical Manual-IV measures change in severity of OCD symptoms from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to starting treatment)
  Interview measure of the presence of OCD, related anxiety disorders and other psychological disorders of childhood.
Clinical Global Impression Severity and Improvement Scales measures change in severity of OCD and co-morbid disorders from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Measure of the severity of the disorders and their improvement as a result of treatment
Global Assessment Scale for Children measures change in overall functioning from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Assesses the overall general functioning of youth under the age of 18.
Child Obsessive-Compulsive Inventory measures change in severity of OCD symptoms from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Assessment of presence of obsessive compulsive symptoms over the past week.
Behavior Rating Inventory of Executive Function measures change in executive functioning from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Neuropsychological measure of executive functioning
Multidimensional Anxiety Scale for Children measures change in severity of anxiety symptoms from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Measure of the presence and severity of anxiety symptoms.
Child Behavior Checklist measures change in severity internalizing and externalizing symptoms from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Broadband measure of child's psychological functioning.
Screen for Child Anxiety and Related Emotional Disorders measures change in severity of anxiety and other disorders from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Measure of the presence and severity of a wide range of emotional disorders.
Brief Symptom Interview measures change in severity of parental psychopathology from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Measure of parental psychopathology
Family Accommodation Scale measures change in parental accommodation from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Measure of the degree to which parents accommodate to their child's OCD.
Test of Everyday Attention-Children's Version measures change in attention from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Neuropsychological measure of the participant's selective, divided, sustained and switching attention
Wisconsin Card Sorting Test Revised and Expanded measures change in executive functioning from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Neuropsychological measure of executive functioning
Delis-Kaplan Executive Function System measures change in executive functioning from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Neuropsychological test of a variety of verbal and nonverbal executive functions.
Children's Color Trails Test measures change in cognitive flexibility from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Neuropsychological test of cognitive flexibility
The Conners' Continuous Performance Test II Version 5measures change in continuous attention from baseline to post-treatment and assesses maintenance of treatment effects at one year and two year follow-up assessments. | Baseline (one week prior to start of treatment, post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Neuropsychological measure of continuous attention.

OTHER OUTCOMES:
Perception of Therapeutic Relationship measures quality of therapeutic relationship at post-treatment and at one year and two year follow-up assessments. | Post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Measure of the participant's perception of the therapeutic relationship
Satisfaction Questionnaire measures satisfaction with treatment at post-treatment and at one year and two year follow-up assessments. | Post treatment (within one week of completing treatment) and follow-ups (six months, and at one year intervals for up to two years following treatment)
  Measures the patient's satisfaction with treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin D. Stark, Ph.D., Principal Investigator — University of Texas
Locations (1):
- Texas Child Study Center, Austin, Texas, United States

REFERENCES:
- See also: Texas Child Study Center — http://www.dellchildrens.net/services_and_programs/texas_child_study_center__mental_health_services/